CLINICAL TRIAL: NCT02019797
Title: Desflurane-induced Myocardial Protection in Aortic Valve Surgery: A Pilot Study
Brief Title: Desflurane-induced Myocardial Protection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nobuyuki Katori (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor-Investigator, Nobuyuki Katori, Assistant Professor, Keio University
Organization: Keio University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Desflurane
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Aortic Valve Stenosis
Keywords: aortic valve replacement
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Desflurane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Desflurane (Experimental): Desflurane inhalation at 1-2 MAC during surgery.
  Interventions: Drug: Desflurane
- Propofol (Active Comparator): 5-8 mg/kg/hr infusion during surgery.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Desflurane — Patients are assigned to desflurane group (Des) or propofol group (Prop). Des receives desflurane (1-2 MAC) inhalation between the induction of anesthesia and before cardiopulmonary bypass (CPB). After the induction of CPB, the anesthesia in Des is switched to a total intravenous anesthesia (TIVA) with propofol. Prop receives a propofol during the surgery.
  Other Names: SUPRANE

SUMMARY:
This study examines pharmacological preconditioning and post conditioning of desflurane by comparing cardiac troponin release in patients receiving either desflurane or propofol for the aortic valve surgery.

DETAILED DESCRIPTION:
Patients scheduled for aortic valve replacement with use of cardiopulmonary bypass are included in the study. Patients are assigned to desflurane group (Des) or propofol group (Prop). Des receives desflurane (1-2 MAC) inhalation between the induction of anesthesia and cardiopulmonary bypass (CPB). After the induction of CPB, the anesthesia in Des is switched to a total intravenous anesthesia (TIVA) with propofol. Prop receives a TIVA during the surgery. All patients receive a continuous infusion of remifentanil. Biomarker of myocardial damage troponin I is examined at 4 points; T1: after the induction of anesthesia, T2: arrival at ICU, T3: 12 hours after the ICU arrival, T4: 24 hours after the ICU arrival, T5: third post operative day (3POD).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for aortic valve replacement with use of cardiopulmonary bypass.

Exclusion Criteria:

* Patients younger than 20 years old.
* Recent myocardial infarction (within 1 year).
* Renal dysfunction (GFR less than 50ml/min).
* Known allergy to study drugs including propofol.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Troponin I | up to 3 days

SECONDARY OUTCOMES:
Length of ICU stay, Length of hospital stay | up to 2 months after the surgery
Acute myocardial infarction | up to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Suematsu, M.D., Ph.D, Study Chair — Keio University
Locations (1):
- Keio University Hospital, Tokyo, Japan